CLINICAL TRIAL: NCT02403310
Title: A Phase 1 Investigator Sponsored Study of Selinexor in Combination With Daunorubicin and Cytarabine in Patients With Previously Untreated Poor-Risk Acute Myeloid Leukemia
Brief Title: A Study of Selinexor in Combination With Daunorubicin and Cytarabine for Untreated AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18157
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Leukemia; Acute Myeloid Leukemia; AML
Keywords: adverse-risk AML; poor-risk karyotype; cytogenetic abnormality; poor-risk mutations; antecedent hematologic disorder; treatment related AML
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Chromosome Aberrations | interventions — selinexor; Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation - Selinexor (Experimental): Dose escalation of selinexor with fixed doses of daunorubicin and cytarabine.
  Induction Therapy may be followed by Consolidation Phase and Maintenance Phase as outlined in the Detailed Description and Intervention Descriptions.
  Interventions: Drug: Selinexor; Drug: Daunorubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: Selinexor — Induction: Oral selinexor on days 1, 3, 8, 10, 15 and 17.
  * Dose Level 2: 80 mg twice weekly.
  * Dose Level 1 (starting dose): 60 mg twice weekly.
  * Dose Level -1: 40 mg twice weekly.
  Consolidation: Selinexor same dose as induction (days 1,3,8,10) unless dose limiting toxicity (DLT) dictates a dose reduction.
  Maintenance: Selinexor at the same dose as induction on days 1 and 8 a 21 day cycle. They will continue for a maximum of 12 months.
  Other Names: KPT-330; SINE KPT-330
Drug: Daunorubicin — Induction: Daunorubicin 60 mg/m^2/day (days 1-3).
  Consolidation: Daunorubicin 45 mg/m^2/day (days 1-2).
  Other Names: Cerubidine®; daunomycin cerubidine; daunorubicin hydrochloride
Drug: Cytarabine — Induction: Cytarabine 100 mg/m^2/day (days 1-7).
  Consolidation: Cytarabine 100 mg/m^2/day (continuous infusion on days 1-5).
  Other Names: Cytosar-U; Tarabine PFS; ARA-C

SUMMARY:
The main purpose of this study is to determine the safety of combining selinexor with daunorubicin and cytarabine. The maximal tolerated dose (MTD) of selinexor with daunorubicin and cytarabine will also be established.

DETAILED DESCRIPTION:
Induction Therapy - Dose escalation of selinexor with Daunorubicin and cytarabine at fixed doses.

Consolidation Phase - Patients who are in complete remission (CR) or complete remission with incomplete count recovery (CRi) by day ≤70 and have recovered from any previous non- hematologic toxicity to baseline or grade ≤1 by day ≤70 following induction chemotherapy may go on to receive consolidation therapy for up to 2 cycles. The consolidation treatment phase will include up to two courses of therapy (28 day cycles) as follows:

Daunorubicin 45mg/m^2/day (days 1-2) Cytarabine 100mg/m^2/day (continuous infusion on days 1-5) Selinexor same dose as induction (days 1,3,8,10) unless dose limiting toxicity (DLT) dictates a dose reduction. Selinexor will be given 2 hours prior to daunorubicin on day 1.

A second cycle of consolidation therapy using the same doses as above will be administered, at the investigators discretion, between 28 and 42 days following initiation of the first consolidation treatment, after peripheral blood counts have recovered to CR, CRi levels, and after recovery from any non-hematologic toxicity to baseline or grade ≤1. Dose escalation of Selinexor will not occur during the consolidation phase.

Maintenance Phase - Patients who remain in CR, CRi after up to 2 cycles of consolidation and are not eligible for allogeneic stem cell transplant will be eligible for the maintenance phase of treatment after recovery from any previous non-hematologic toxicity to baseline or grade ≤1. Maintenance therapy will consist of:

Selinexor at the same dose as induction on days 1 and 8 of a 21 day cycle. They will continue for a maximum of 12 months.

Expansion Phase - Once the MTD has been established, there will be an expansion phase to enroll an additional 13 subjects at the MTD to better characterize the safety profile and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants must have newly diagnosed, previously untreated acute myeloid leukemia (AML) (excluding M3); Must have adverse-risk AML defined as poor-risk karyotype (complex, monosomal or other known poor risk cytogenetic abnormality), poor-risk mutations/fusion genes or known history of antecedent hematologic disorder, or treatment related AML, or be ≥60 years of age; Cytogenetics, FISH or mutational analysis confirming adverse risk features must have been done within 90 days prior to enrollment.
* May not have undergone any prior therapy for their AML other than hydroxyurea. However, if patients had an antecedent myelodysplastic syndrome (MDS), prior treatment with a hypomethylating agent or any other therapy (with the exception of allogeneic stem cell transplant) used to treat their MDS is allowed.
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Life expectancy of greater than 2 months
* Must have normal organ function
* Able and willing to adhere to the study visit schedule and other protocol requirements
* Baseline left ventricular ejection fraction (LVEF) ≥ 50%
* Women of child-bearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 50 milli-international units per milliliter (mIU)mL) within 10 days and again within 24 hours prior to beginning study treatment. Participants of childbearing potential must practice recommended contraception. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Breastfeeding mothers must agree to discontinue nursing if the mother is treated with selinexor.
* Ability to understand and the willingness to sign a written informed consent document
* Able to swallow capsules and have no evidence of GI tract abnormality that would alter the absorption of oral medications
* Prothrombin time (PT) and partial thromboplastin time (PTT) ≤ 1.5 x upper limit of normal (ULN)

Exclusion Criteria:

* May not be receiving any other investigational agents
* Documented central nervous system (CNS) involvement of AML
* AML with favorable risk cytogenetic abnormalities including t(15;17), t(8;21) or inv(16)
* Potential participants who are in the blast phase of chronic myeloid leukemia
* Major surgery within 2 weeks of first dose of study drug; must have recovered from the effects of any surgery performed greater than 2 weeks prior
* White blood cell (WBC) count ≥50,000 on hydroxyurea
* Predicted inability to tolerate standard induction chemotherapy with daunorubicin and cytarabine
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* HIV-positive, receiving combination anti-retroviral therapy
* No other malignancies in addition to AML that are currently requiring treatment with the exception of basal cell or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast
* History of allogeneic stem cell transplant for MDS or any other antecedent hematologic disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-06-18 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Maximal Tolerated Dose (MTD) of Selinexor | Up to 18 months
  MTD / Recommended Phase II Dose (RP2D) of selinexor with daunorubicin and cytarabine. Dose Limiting Toxicity (DLT): Non-hematologic - Any grade 3-4 drug-related non-hematologic toxicity, with the following exceptions: Nausea/vomiting or diarrhea adequately controlled with antiemetics/antidiarrheals; Infection or febrile neutropenia adequately controlled with antibiotics; Liver function abnormalities (without clinical symptoms) that recover to baseline or grade 0-1 within 7 days; Grade 3-4 electrolyte or metabolic laboratory abnormalities that are not considered clinically significant by the treating investigator/physician and that recover to baseline or grade 0-1 within 7 days; Alopecia. Hematologic - Grade 3-4 neutropenia and/or thrombocytopenia (thought to be due to marrow hypoplasia and NOT leukemic burden) that does not recover to grade ≤2 by day 56.

SECONDARY OUTCOMES:
Rate of Complete Response (CR) Plus Complete Response with Incomplete Count Recovery (CRi). | Up to 18 months
  A CR designation requires that the patient achieve the morphologic leukemia-free state and have an absolute neutrophil count of more than 1,000/μL and platelets of 100,000/μL. A CRi designation requires that the patient achieve the morphologic leukemia-free state with incomplete recovery of neutrophils (<1,000/μL) or platelets (<100,000/μL).
Disease Free Survival (DFS) | Up to 18 months
  Disease free survival is measured from the time measurement criteria are met for CR/CRi until the first date that relapse is objectively documented.
Time to Progression (TTP) | Up to 18 months
  Time to progression is a secondary endpoint that will be measured as the time from when the patient started treatment to the time the patient is first recorded as having relapsed, or the date of death if the patient dies due to causes other than disease progression.
Overall Survival (OS) | Up to 18 months
  Overall survival is a secondary endpoint that will be measured as time from the start of treatment until death from any cause, or the last date the patient was known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Kendra Sweet, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States